CLINICAL TRIAL: NCT01577992
Title: Evaluation of the Subjective and Objective Painful Threshold in Multiple System Atrophy Pain and Multiple System Atrophy
Acronym: MSA-DOUL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0931403; HAO 2009 (Other: CHU de Toulouse)
Record Dates: First submitted 2011-11-07; First posted 2012-04-16 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Pain Threshold; Multiple System Atrophy
Keywords: subjective pain; Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: MSA disease (Experimental): determination of objective and subjective pain threshold before and after levodopa intake
  Interventions: Drug: Levodopa test
- Group 2: Parkinson disease (Experimental): determination of objective and subjective pain threshold before and after levodopa intake
  Interventions: Drug: Levodopa test
- Group 3: healthy volunteers. (Other): one determination of objective and subjective pain threshold without treatment
  Interventions: Procedure: determination of objective and subjective pain threshold

INTERVENTIONS:
Drug: Levodopa test — Each patients with PD and MSA will be evaluated in two conditions : OFF (without dopaminergic treatment since 12h) and ON condition (after a L-DOPA dose. This dose will be 150% of the DOPA morning dose. The healthy volunteers will be evaluated in only one condition (without L-DOPA administration)
  Arms: Group 1: MSA disease; Group 2: Parkinson disease
Procedure: determination of objective and subjective pain threshold — Test without levodopa intake
  Arms: Group 3: healthy volunteers.

SUMMARY:
Multiple system atrophy (MSA) is a sporadic neurodegenerative disorder. MSA is dominated by autonomic/urogenital failure which may be associated with either Parkinsonism (MSA-P subtype) or with cerebellar ataxia (MSA-C subtype). The prognostic of this disease is bad because it ended with the patient's death few years later. No neuroprotective treatment has shown a real efficacy. 50% of patients suffering of MSA frequently experienced painful sensation. The origin of this pain is unknown. In Parkinson disease (PD) ; arguments suggest the implication of dopamine neuromediator pathway in integration and modulation of pain. Several studies suggest the existence of various influences with dopamine implication in the appearance of painful sensation and that would be inhibitory. That's why observed painful symptoms in MSA and PD could be due to a decrease of pain appearance threshold, secondary to a lost of control of sensitizes centres, to Parkinson control.

It is interesting to determine if MSA as PD is responsible for a decrease of pain threshold and to characterise the levodopa effect on the patient's pain threshold. Better physiopathology knowledge of pain in MSA is necessary to improve the therapeutic care. Because the efficacy of others treatments is low, it's important to improve the research for a better comfort of patients with a better understanding, analysing and treating of the pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 50 to 80 years old (Male and female)
* Patients suffering of a diagnosis possible or probable MSA-P with the international criteria (2008).
* Patients with clinical diagnosis of Parkinson's disease according to the criteria of the UKPDSBB (Gibb et Lees, 1988; Hughes et al, 1992)
* Patients with no cognitive troubles
* Patients who give their informed and signed consent.
* Patients affiliated to a social protection program

Exclusion Criteria:

* Patient suffering from an other parkinson syndrome than MSA and PD, by example progressive supranuclear palsy, corticobasal degeneration…
* Patient suffering of a diagnosis possible or probable MSA-C with the international criteria
* Patient suffering from another pathology causing chronic pain (rheumatic disease, traumatic or orthopedic pathologies…)
* Patient under tutelage, curatella or law protection

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Subjective pain threshold | 60 minutes
  Subjective pain threshold determined using thermal stimulation (Thermotest) with the method of levels, before and after levodopa intake for MSA patients and PD patients and once for healthy volunteers

SECONDARY OUTCOMES:
Objective nociceptive pain threshold | 15 minutes
  Objective nociceptive pain threshold thanks to reflex of flexion (reflex RIII)before and after levodopa intake for MSA patients and PD patients and once for healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Christine Brefel-Courbon, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, neurology, Toulouse, France